CLINICAL TRIAL: NCT03579147
Title: Safety and Patient Satisfaction With Noninvasive Repetitive Pulse Magnetic Stimulation (rPMS) for Aesthetic Improvements of Buttocks
Brief Title: Non-invasive Buttock Lifting Induced by Magnetic Device - Multicentric Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It was not possible to recruit any patients at that time.
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-Buttocks_001
Record Dates: First submitted 2018-06-19; First posted 2018-07-06 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Muscle Tightness
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment Group (Experimental): Treatment with the investigational device BTL EMSCULPT.
  Interventions: Device: Treatment with BTL EMSCULPT device

INTERVENTIONS:
Device: Treatment with BTL EMSCULPT device — The treatment administration phase will consist of four (4) treatments, delivered twice a week. The applicator will be applied over the buttock area. Visible contractions will be induced by the device.

SUMMARY:
This study will evaluate the clinical safety and patient satisfaction with the high power magnet system for the aesthetic improvement of buttocks. The study is a prospective multi-center open-label single-arm study. The subjects will be enrolled and assigned into a single study group. Subjects will be required to complete four (4) treatment visits and three follow-up visits - 1 month, 3 months and 12 months after the final treatment. Study will be conducted at several study sites.

At the baseline visit, subject's weight will be recorded. Subjects will receive Buttocks Evaluation Questionnaire to fill in.

The treatment administration phase will consist of four (4) treatments, delivered twice a week. The applicator will be applied over the gluteal area. Visible contractions will be induced by the device.

At the last therapy visit, the subject's weight will be recorded. In addition, subjects will receive Subject Satisfaction, Buttocks Evaluation and Therapy Comfort Questionnaires to fill in.

Safety measures will include documentation of adverse events (AE) including subject's experience of pain or discomfort after the procedure. Following each treatment administration and at the follow-up visits, subjects will be checked for immediate post-procedure adverse event assessment.

Post-procedure evaluation (follow-up visits) will be conducted 1 month, 3 months and 12 months after the final treatment. A weight measure will be conducted. Also, subject's satisfaction and buttocks evaluation will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed informed consent form
* BMI ≤ 30 kg/m2
* Women of child-bearing potential are required to use birth control measures during the
* whole duration of the study
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring during study participation
* Subjects willing and able to maintain his/her regular (pre-procedure) diet and exercise regimen without effecting significant change in either direction during study participation

Exclusion Criteria:

* Cardiac pacemakers
* Electronic implants
* Pulmonary insufficiency
* Metal implants
* Drug pumps
* Haemorrhagic conditions
* Anticoagulation therapy
* Heart disorders
* Malignant tumor
* Fever
* Pregnancy
* Breastfeeding
* Following recent surgical procedures when muscle contraction may disrupt the healing process
* Application over menstruating uterus
* Application over areas of the skin which lack normal sensation
* Scars, open lesions and wounds at the treatment area
* Unrepaired abdominal hernia

Min Age: 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Subject's satisfaction | 13 months
  The 5-point Likert scale Subject Satisfaction Questionnaire will be used for an analysis of the subject's opinion of the therapy results. Subjects will be evaluating agreement with three different statements (concerning satisfaction with therapy results and appearance of abdominal area after therapy) by choosing an answer on a scale between 1 (Strongly disagree) and 5 (Strongly agree). Minimally 80% of the treated subjects should report the agreement with all three statements given in the questionnaire (answers "Agree" and "Strongly agree") in order to claim subject's satisfaction with the therapy outcome.
Effectiveness of the device assessed through Buttocks Evaluation Questionnaire | 13 months
  The 7 point Likert scale Buttocks Evaluation Questionnaire will be used for an assessment if there is a change in subject's perception of their own buttocks area before and after the therapy session. The total possible score ranges from 4 points (lowest possible satisfaction) to 28 points (highest possible satisfaction).

SECONDARY OUTCOMES:
Occurrence of treatment-related adverse events | 13 months
  The secondary objective of the study is to determine side effects and adverse events (AE) associated with the treatment of the abdominal area.
  The occurrence of adverse events will be followed throughout the whole study.
Therapy comfort | 3 months
  Therapy comfort will be noted at the last therapy visit. Subjects will be asked to evaluate the agreement with the statement concerning the conformity of the study treatment. Subjects will be evaluating the agreement by choosing an answer on a scale between 1 (Strongly disagree) and 5 (Strongly agree). Based on a given answers, the therapy comfort will be calculated.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - Contour Medical, Gilbert, Arizona
  - Plastic Surgery Excellence, Beverly Hills, California
  - Dr. Mariano Busso Aesthetic Dermatology, Miami, Florida
  - Chicago Cosmetic Surgery and Dermatology, Chicago, Illinois
  - Ovation Med Spa, Houston, Texas
  - Refresh Dermatology, Houston, Texas
- Aesthe Clinic, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No